CLINICAL TRIAL: NCT01425060
Title: Improving Effective Contraceptive Use Among Opioid-maintained Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Sarah Heil, Associate Professor of Psychiatry and Psychology, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34DA030534 (NIH)
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Contraceptive Usage; Opioid Dependence
Keywords: Contraception; Unintended pregnancy; HIV; HIV Risk; Sexually Transmitted Infections; Women; Pregnancy; Neonatal Health; Drug Use; Drug Treatment; Opioids
MeSH Terms: conditions — Contraception Behavior; Opioid-Related Disorders; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Contraceptive management program (Experimental)
  Interventions: Behavioral: Contraceptive management program
- Usual care (Active Comparator): The usual care condition will be given general information about contraceptive options and contact information for clinics and providers that provide contraceptive services.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Contraceptive management program — The contraceptive management program will consist of two components: (1) the World Health Organization's contraception protocol and (2) reinforced follow-up visits.
  Arms: Contraceptive management program
Other: Usual care — The usual care condition will be given general information about contraceptive options and contact information for clinics and providers that provide contraceptive services.
  Arms: Usual care

SUMMARY:
Nearly 9 of every 10 pregnant opioid-dependent women report that the current pregnancy was unintended and the majority of non-pregnant opioid-maintained women do not use contraception or use less effective methods like condoms. This proposal aims to develop and test a novel contraceptive management program to increase use of more effective contraceptives among opioid-maintained women and to examine the impact of more effective contraceptive use on condom use. The proposed research may reduce unintended pregnancy among opioid-dependent women without increasing their risk of sexually transmitted infections and the knowledge gained will also have implications for addressing high rates of unintended pregnancy in the general population.

DETAILED DESCRIPTION:
The rate of unintended pregnancy among opioid-dependent women is extremely high: nearly 9 of every 10 pregnant opioid-dependent women report that the current pregnancy was unintended, a rate 2-3 times that of the general population. Despite these dire statistics, there is a dearth of scientific knowledge about contraceptive use in this population and about how to promote use of more effective contraceptives (e.g., birth control pills, IUDs, implants).

The aim of this Stage I Behavioral and Integrative Treatment Development Program application is to develop and pilot test a novel contraceptive management program to increase use of more effective contraceptives among OM women. OM women (N=100) at risk for unintended pregnancy will be randomly assigned to a 6-month contraceptive management program or to usual care. The contraceptive management program will consist of two components: (1) the World Health Organization's contraception protocol and (2) reinforced follow-up visits. At their first visit, participants assigned to the contraceptive management program will complete the WHO's contraception protocol, which consists of assistance choosing a contraceptive method, structured educational counseling about their chosen method, a free supply of this method, and the option of initiating this method immediately. Subsequently, contraceptive management program participants will earn voucher-based incentives to reinforce attendance at follow-up visits where they will receive support to manage side effects and problem-solve compliance problems, refills of their chosen method, and assistance switching methods when indicated. At each visit, contraceptive management program participants will also be counseled about the risks of sexually transmitted infections (STIs), including HIV/AIDS, the need for dual protection (i.e., protection from both pregnancy and STIs), and provided with a supply of condoms. Participants assigned to the usual care condition will be given general information about contraceptive options and contact information for clinics and providers that provide contraceptive services. Contraceptive use by all participants will be evaluated at assessments scheduled 1, 3, and 6 months after trial intake. The impact of prescription contraceptive use on condom use will also be assessed. It is hypothesized that the contraceptive management program will increase effective contraceptive use without decreasing condom use.

The proposed project will be the seminal study of an intervention to increase more effective contraceptive use in OM women and the first step towards our overarching goal of developing an efficacious, empirically based contraceptive management program that can be disseminated to drug treatment facilities throughout the country. The proposed research also holds significant potential for impacting public health in general, as development of efficacious programs will help reduce the vast economic and societal costs associated with unintended pregnancy among drug-dependent and non-drug-dependent women alike.

ELIGIBILITY:
Inclusion Criteria:

* 18-44 years of age
* pre-menopausal and have no history of a tubal ligation or hysterectomy
* have had heterosexual vaginal sex in the past 12 months
* have no plans to become pregnant in the next 6 months
* be medically eligible to use prescription contraceptives
* report no prescription contraceptive method use (i.e., no use of pills, patch, ring in the past 7 days or depot injections, implants, or IUD in the past 3 months) OR report primary use of a non-prescription method (i.e., condoms, sponge, diaphragm, withdrawal, or rhythm method)
* have been in opioid maintenance treatment for at least the past 30 days
* be English-speaking.

Exclusion Criteria:

* failure to meet the aforementioned inclusion criteria
* refusal to participate

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Point prevalence use of a prescription contraceptive | 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Sarah H. Heil, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont Substance Abuse Treatment Center, Burlington, Vermont, United States

REFERENCES:
- [Background] Heil SH, Higgins ST. The scientific and ethical rationale for using incentives to promote contraceptive use among drug-abusing women. Addiction. 2012 Jun;107(6):1044-6. doi: 10.1111/j.1360-0443.2012.03798.x. No abstract available. PMID 22563830
- [Background] Heil SH, Gaalema DE, Johnston AM, Sigmon SC, Badger GJ, Higgins ST. Infant pupillary response to methadone administration during treatment for neonatal abstinence syndrome: a feasibility study. Drug Alcohol Depend. 2012 Nov 1;126(1-2):268-71. doi: 10.1016/j.drugalcdep.2012.05.006. Epub 2012 Jun 8. PMID 22682657
- [Background] Hand DJ, Heil SH, Sigmon SC, Higgins ST. Improving medicaid health incentives programs: lessons from substance abuse treatment research. Prev Med. 2014 Jun;63:87-9. doi: 10.1016/j.ypmed.2014.03.001. Epub 2014 Mar 12. PMID 24613792
- [Background] Herrmann ES, Hand DJ, Johnson MW, Badger GJ, Heil SH. Examining delay discounting of condom-protected sex among opioid-dependent women and non-drug-using control women. Drug Alcohol Depend. 2014 Nov 1;144:53-60. doi: 10.1016/j.drugalcdep.2014.07.026. Epub 2014 Jul 30. PMID 25190049
- [Background] Meyer MC, Johnston AM, Crocker AM, Heil SH. Methadone and buprenorphine for opioid dependence during pregnancy: a retrospective cohort study. J Addict Med. 2015 Mar-Apr;9(2):81-6. doi: 10.1097/ADM.0000000000000092. PMID 25622120